CLINICAL TRIAL: NCT04760743
Title: A Phase I, Placebo-controlled, Randomized, Observer-blinded, Dose-escalation Study to Assess the Safety, Reactogenicity, and Immunogenicity of a SARS-CoV-2 Vaccine (NBP2001) in Healthy Adults Aged at 19 to 55 Years
Brief Title: Safety and Immunogenicity of a SARS-CoV-2 Vaccine (NBP2001) in Healthy Adults (COVID-19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NBP2001_001
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 (Healthy Volunteers)
MeSH Terms: conditions — COVID-19 | interventions — aluminum sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose level cohort (Experimental): 2 dose of NBP2001 adjuvanted with alum (Receptor Binding domain (RBD) 30μg/dose), 1 dose each on Day 0 and 28
  Interventions: Biological: NBP2001 adjuvanted with alum (RBD 30μg/dose)
- high dose level cohort (Experimental): 2 dose of NBP2001 adjuvanted with alum (Receptor Binding domain (RBD) 50μg/dose), 1 dose each on Day 0 and 28
  Interventions: Biological: NBP2001 adjuvanted with alum (RBD 50μg/dose)
- Placebo group (Placebo Comparator): 2 doses of Placebo Saline, 1 dose each on Days 0 and 28.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: NBP2001 adjuvanted with alum (RBD 30μg/dose) — Participants will receive intramuscular (IM) injections of NBP2001(RBD 30μg/dose) on Days 0 and 28.
  Arms: low dose level cohort
Biological: NBP2001 adjuvanted with alum (RBD 50μg/dose) — Participants will receive intramuscular (IM) injections of NBP2001(RBD 50μg/dose) on Days 0 and 28.
  Arms: high dose level cohort
Other: Normal Saline — Participants will receive intramuscular (IM) injections of Normal saline on Days 0 and 28.
  Arms: Placebo group

SUMMARY:
This study is to assess the safety, reactogenicity and immunogenicity of a SK SARS-CoV-2 recombinant protein subunit vaccine (NBP2001) in healthy adults.

DETAILED DESCRIPTION:
This is a first-in-human, Phase I, randomized, placebo-controlled, observer-blinded study to assess the safety, reactogenicity and immunogenicity of a SK SARS-CoV-2 recombinant protein subunit vaccine (NBP2001) in healthy adults.

A total of 50 healthy adults between 19 and 55 years of age will be enrolled and block-randomized in a 4:1 ratio to receive 2 doses of either one NBP2001 formulation (Test group 1 or 2) or placebo saline (Placebo group).

Over the study period, participants will commonly attend 10 planned visits. Telephone calls will be made 7 days after each vaccination (Day 7+3 after Visit 2 and Visit 4). However, sentinel participants will be required to return at Day 7(+ 3 days) after 1st vaccination for rigorous safety assessment.

Study vaccination will comprise 2 intramuscular injections of saline placebo, or a 30 or 50μg dose of NBP2001 in an injection volume of approximately 0.5mL. The study vaccines will be injected preferably into the deltoid muscle of the upper arm at a 28-day interval.

Halting rules based on reactogenicity and safety outcomes are defined, and enrollment and study vaccination may be paused during the study if any halting rules are met.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant must be 19 to 55 years of age inclusive, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Participants who are healthy as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, and medical judgement of the investigator
3. Participants who are able to attend all scheduled visits and comply with all study procedures.

   Weight
4. Body mass index (BMI) within the range 18-30 kg/m2 at screening (inclusive)

   Sex and Contraceptive/Barrier Requirements
5. Female participants of childbearing potential must agree to be heterosexually inactive, or agree to consistently use at least one acceptable method of contraception from at least 21 days prior to the 1st study vaccination to 8 weeks after the last study vaccination
6. Female participants with a negative urine or serum pregnancy test at screening

   Informed Consent
7. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Medical Conditions

1. Any clinically significant respiratory symptoms (e.g. cough, sore throat), febrile illness (tympanic temperature >38°C), or acute illness within 72 hours prior to the 1st study vaccination. A prospective participant should not be included until 72 hours after the condition has resolved.
2. History of virologically-confirmed COVID-19 disease, or definite or suspected exposure to anyone known to have SARS-CoV-2 infection
3. History of virologically-confirmed SARS or MERS disease
4. History of congenital, hereditary, acquired immunodeficiency, or autoimmune disease
5. Any positive test results for hepatitis B, C, or HIV at screening
6. History of bleeding disorder or thrombocytopenia which is contraindicating intramuscular vaccination in the investigator's opinion
7. History of hypersensitivity and severe allergic reaction (e.g. anaphylaxis, Guillain-Barre syndrome) to any vaccines or components of the study intervention
8. History of malignancy within 5 years prior to the 1st study vaccination
9. Significant chronic illness that, in the opinion of the investigator, might increase risk of severe COVID-19, or interfere with the evaluation of the study objectives (e.g. asthma, chronic pulmonary disease, cardiovascular disease, chronic liver disease, diabetes mellitus, uncontrolled hypertension, renal disorders)
10. History of, or planned surgery under general anesthesia from 1 year prior to the 1st study vaccination through the study period
11. Any other conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives (e.g. neurologic or psychiatric conditions)
12. Female participants who are pregnant or breastfeeding
13. Current smokers or a recent smoking history within 12 weeks prior to the 1st study vaccination. Occasional smokers who smoke up to 10 cigarettes per month may be allowed to participate at the investigator's discretion

    Prior/Concomitant therapy
14. Receipt of any medications or vaccinations intended to prevent COVID-19.
15. Receipt of any vaccine within 4 weeks prior to the 1st study vaccination or planned receipt of any vaccine from enrollment through 28 days after the last study vaccination (Visit 7), except for influenza vaccination, which may be received at least 2 weeks prior to the 1st study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines
16. Receipt of immunoglobulins and/or any blood or blood products within 12 weeks prior to the 1st study vaccination
17. Chronic use (more than 2 consecutive weeks) of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (≥10mg prednisone/day or equivalent for more than 2 consecutive weeks) within 12 weeks prior to the 1st vaccination. The use of topical and nasal glucocorticoids will be permitted.

    Prior/Concurrent Clinical Study Experience
18. Participation in another clinical study involving study intervention within 6 months prior to the 1st study vaccination, or concurrent, planned participation in another clinical study with study intervention during this study period.

    Other Exclusions
19. Investigators, or study staff who are directly involved in the conduct of this study or supervised by the investigator, and their respective family members.
20. Healthcare worker or emergency response personnel in an occupation with a high risk of exposure to SARS-CoV-2

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of immediate systemic reactions | Through 30 minutes (2 hours for sentinel participants) post-vaccination
Occurrence of solicited local Adverse Events (AEs) during 7 days post each vaccination | Through 7 days post-vaccination
Occurrence of solicited systemic AEs during 7 days post each vaccination | Through 7 days post-vaccination
Occurrence of unsolicited AEs during 28 days post each vaccination | Through 28 days post-vaccination
Occurrence of Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs) and Adverse Events of Special Interest (AESIs) during the whole study period | Through Day 0 to Day 365 post last vaccination
GMT of IgG antibody to the SARS-CoV-2 RBD measured by Enzyme-linked Immunosorbent Assay (ELISA) | Through Day 365 post last vaccination
GMFR of IgG antibody to the SARS-CoV-2 RBD from baseline measured by ELISA | Through Day 365 post last vaccination
Percentage of participants with ≥ 4-fold rise from baseline in ELISA IgG titer | Through Day 365 post last vaccination
GMT of neutralizing antibody to the SARS-CoV-2 measured by pseudovirus and wild-type virus neutralization assays | Through Day 365 post last vaccination
GMFR of neutralizing antibody to the SARS-CoV-2 from baseline measured by pseudovirus and wild-type virus neutralization assays | Through Day 365 post last vaccination
Percentage of participants with ≥ 4-fold rise from baseline in pseudovirus and wild-type neutralizing antibody titer | Through Day 365 post last vaccination
Cell-mediated response for both Th1 and Th2 (e.g. INF-γ, IL-4 using Enzyme-linked ImmunoSpot (ELISpot) or other system | Through Day 28 post last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Myoung-Don Oh, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Bundang
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No